CCR no: 5287 IRAS no: 282755

Version Date: 10th July 2020

**Version Number: 2.0** 

## The ROYAL MARSDEN NHS Foundation Trust

GI & Lymphoma Unit Fulham Road, London SW3 6JJ: 020-7808-2153 Downs Road, Sutton SM2 5PT: 020-8661-3156

> The Royal Marsden Downs Road, Sutton Surrey SM2 5PT Tel: 02086426011 www.royalmarsden.nhs.uk

#### PATIENT INFORMATION SHEET

#### **CARDS**

# Cancer: Rapid Diagnostics and Immune assessment for SARS-CoV-2 (COVID-19) ARM A

We invite you to take part in a research study. Before deciding whether to take part, it is important that you understand why the research is being done and what it will involve. Please take time to read this carefully and discuss it with other people if you wish. Please ask your doctor or nurse if there is anything you do not understand or if you want more information. Please take your time to decide.

#### Why am I being invited to take part in this study?

Your doctor has invited you to take part in this study because you are having or have had tests of suspected Coronavirus (COVID-19) infection which is caused by a virus named SARS-CoV-2. We would like to be able to collect information on your medical condition, and collect additional blood, saliva and throat/nose swab samples from you and/or during each of your subsequent visits to hospital.

If the throat/nose swab confirms you have COVID-19 infection, or if your doctor believes you have COVID-19 despite a negative test, we would like to use these additional samples for our research project, which is described in detail below. If you do not have COVID-19 infection, we would not collect any further clinical information or samples for the purposes of our study.

#### What is the purpose of this study?

Infection caused by COVID-19 has been responsible for a large number of deaths in the UK and around the world.

People who are receiving therapy for cancer sometimes have a lowered immune system. In this project, we want to study the effect of COVID-19 infection in people with cancer. We are

CCR no: 5287 IRAS no: 282755

Version Date: 10th July 2020


investigating the effect of COVID-19 infection in people with cancer. We will study your body's immune system and its response to the COVID-19 virus.

You will be helping us to find out:

- 1. Whether people with cancer have different symptoms of COVID-19
- 2. How your body develops immunity to the virus
- 3. How long it takes your body to clear the virus
- 4. How cancer treatments can be safely started after COVID-19
- 5. If we can develop a much quicker and accurate test for the COVID-19 virus which would enable rapid identification of people infected with the virus so that we will be able to treat them more quickly.

#### What will happen to me if I take part?

If you agree to take part in this study, any tests or treatment that your doctor recommends for you will not be affected by your taking part in this study. Up to 4 extra visits to the hospital will be necessary for the purpose of this study. Visits will take approximately 15-20 minutes. Where possible, some of these visits will be incorporated into your pre-existing hospital appointments.

- We are asking for your permission to collect information about your medical history, cancer and previous treatments at the Royal Marsden Hospital (RM). We will collect this information from your medical records. We are also asking for your permission to contact your GP to obtain updated information. All of the information we collect will be anonymised at this stage so that researchers will not be able to identify you from the data collected. The majority of the work carried out on your samples will be conducted at the Royal Marsden Hospital and St George's Hospital but we may also on occasion share your anonymised information with other national or international institutions with whom we collaborate in ethically approved studies.
- We are asking for your permission to take additional saliva, blood and throat/nose swabs samples when you are investigated for COVID-19 infection. We would like to take two swabs from your throat/nose (one of which you would have as part of your standard testing for COVID-19 infection regardless of whether or not you decide to take part in the study), a blood sample of no more than 30 mL (about 6 teaspoons) and a saliva sample.
- If you have COVID-19, we would like to take more blood, saliva, and throat/nose swabs in 7\* 14, 28, 42 and 56 days. \*Day 7 samples are only required if you are an inpatient at the Royal Marsden Hospital.
- We are asking for your permission to perform research on the swabs, saliva and blood samples.
- If your COVID-19 test is negative, and your doctor believes you do not have COVID-19 you
  will no longer be involved in the study and any samples taken for research purposes will be
  disposed of. You could be reconsidered for the study if you develop new symptoms of
  COVID-19 infection.

CCR no: 5287 IRAS no: 282755

Version Date: 10th July 2020


Once you have read this information sheet and signed the consent form, we will start collecting clinical information in an anonymised fashion and we will inform your GP. If you have given your consent, we will arrange for research blood, saliva, throat/nose swab samples to be taken. All samples will also be anonymised.

All of the anonymised samples will be collected at the Royal Marsden Hospital, and will be sent to and stored at St Georges Hospital where the appropriate analyses will be performed. These researchers will not be able to identify you. You should be aware that the scientists might not conduct all research immediately, but that your samples may be studied at a later point in time.

### What will happen if I lose capacity to consent during the study or I don't want to carry on with the study?

If you decide to take part, and later change your mind, you are free to withdraw your permission. You do not have to give a reason for your decision and this will have no influence over your future medical care. After withdrawing consent no samples will be collected or any research procedure carried out. You will be given the option of whether further data can be collected and whether the samples you have already contributed can continue to be used in research. The data collected about you up until the point of withdrawal of consent will still be used in the data analysis for the study.

What is capacity and loss of capacity? Capacity means the ability to use and understand information to make a decision, and communicate any decision made. A person lacks capacity if their mind is impaired or disturbed in some way, which means they're unable to make a decision at that time.

In the event that you lose capacity we will ask for further consent from your designated personal consultee. In the event that your personal consultee is unavailable or cannot be reached we will seek advice from a nominated consultee, who is a person independent of the project appointed in accordance with the Department of Health's guidance. When you regain capacity, we will ask for your consent again.

#### What are the possible risks and benefits of taking part?

#### Benefits

Information that we will obtain from your samples will not affect the way you will be treated, and you will not be informed of the results. There will be no direct benefit to you from your participation in this study. We are asking for your permission to study and store your samples now and in the future (indefinitely) at the Royal Marsden Hospital, St Georges Hospital, and other approved offsite facilities. These samples may be used in other ethically approved COVID-19 studies. The analysis of the samples you provide during this study may help us develop understanding and tests that will improve the treatment of people with cancer in the future.

#### Risks associated with taking blood

Risks associated with taking blood from a vein in your arm include pain, bruising, light-headedness and on rare occasions, infection.

Risks associated with throat/nose swabs

CCR no: 5287 IRAS no: 282755

Version Date: 10th July 2020


There may be a small amount of discomfort within the throat/nose.

Risks associated with collection of saliva

There are not thought to be any particular risks associated with providing a saliva sample.

Sometimes these types of samples can help to establish products that could be patented and licensed. Your samples would be considered a donation, and you would not benefit financially. Research carried out at our Institution is not for commercial purposes, but to help us understand how to improve the clinical management of COVID-19 infection in people with cancer.

If you have private medical insurance, please check with the company before agreeing to take part to ensure that your medical insurance will not be affected. Neither you nor your doctor will be told of the results of the additional research tests.

#### Will I be reimbursed for participating in this study?

We would be extremely grateful for your participation in this study. You will be entitled to free parking\* for any visits to hospital for the study. You will not receive any payment for participating in this study. Similarly, other costs of transport (e.g. fuel, public transport) will not be reimbursed. \*If you require parking, please discuss this with your Research Nurse/Research team member prior to your study visit.

#### What if something goes wrong?

If you have any concerns about this study you should speak to your research doctor/nurse who will do their best to answer your questions. If you are harmed by taking part in this research project, there are no special compensation arrangements. Healthcare professionals working on clinical trials are covered by NHS Indemnity and if you are harmed due to someone else's negligence, you may have grounds for legal action but you may have to pay for it. If you wish to complain about any aspect of the way you have been approached or treated during the course of this study, the National Health Service complaints mechanisms will be available to you. Concerns should be raised by speaking to a member of staff at your hospital or by talking to the local Patient Advice and Liaison Service (PALS) which has been established in every NHS trust. Contact details can be found towards the end of this patient information sheet.

#### Will my taking part in this study be kept confidential?

All the information which is collected about you will be kept strictly confidential. Your blood, saliva, and throat/nose swab samples for research will be anonymised so that researchers will not be able to identify you. A unique subject identifier will be allocated to you which will be used to label your data and samples which is only accessible to the research team at the Royal Marsden Hospital. Regulatory authorities, monitors and auditors may have access to personal identifiable data. Any information about you or about the result of the research tests will be kept confidential and will not be included in your medical records.

In this research study we will use information from you, your medical records and possibly your GP. We will only use information that we need for the research study. We will let very few people know your name or contact details, and only if they really need it for this study.

CCR no: 5287 IRAS no: 282755

Version Date: 10th July 2020


Everyone involved in this study will keep your data safe and secure. We will also follow all privacy rules. At the end of the study we will save some of the data in case we need to check it and for future research. We will make sure no-one can work out who you are from the reports we write.

#### What will happen to the results of the research study?

The results are likely to be published in a medical journal or presented at a medical conference. However, you will not be identified in any report or publication produced from this study. When the study is completed, we aim to make the results available to view on a clinical trials database (<a href="https://clinicaltrials.gov">https://clinicaltrials.gov</a>). If you do not have access to a computer and would like to know the results, please get in touch with the trial team who can arrange to send you or your family a copy.

#### Who is organising the research?

This research is sponsored by the Royal Marsden NHS Trust. Your doctor will not receive any personal financial payment if you take part.

#### Who reviewed the study?

This study has been approved by a Committee for Clinical Research (CCR), Health Research Authority (HRA) and Research Ethics Committee (REC) on behalf of hospitals throughout the UK.

#### What happens now?

Your doctor or nurse will be happy to answer any questions you may have regarding the study. Once you have read and understood the information contained in this patient information sheet and your questions have been answered you will be asked to decide whether you want to participate in this study. Additional research samples will be obtained at the same time as your standard diagnostic test and so you will need to make a decision prior to this being collected. Once you have reached your decision, please inform your doctor or nurse.

#### **General Data Protection Regulation (GDPR) Transparency Statement**

#### How will we use information about you?

We will need to use information from you, your medical records and possibly your GP for this research project.

This information will include your

- Name/Initials
- · Date of birth
- Hospital number
- NHS Number
- Contact details

People will use this information to do the research or to check your records to make sure that the research is being done properly.

CCR no: 5287 IRAS no: 282755

Version Date: 10th July 2020


People who do not need to know who you are will not be able to see your name or contact details. Your data will have a code number instead.

We will keep all information about you safe and secure.

Once we have finished the study, we will keep some of the data so we can check the results. RM will keep identifiable information about you for at least 5 years after the study has finished, in line with local policies and legal requirements. We will write our reports in a way that no-one can work out that you took part in the study.

#### What are your choices about how your information is used?

- You can stop being part of the study at any time, without giving a reason, but we will keep information about you that we already have.
- If you choose to stop taking part in the study, we would like to continue collecting information about your health from the Royal Marsden Hospital and your GP. If you do not want this to happen, tell us and we will stop.
- We need to manage your records in specific ways for the research to be reliable. This means that we won't be able to let you see or change the data we hold about you.
- If you agree to take part in this study, you will have the option to take part in future research using your data saved from this study.

#### Where can you find out more about how your information is used?

You can find out more about how we use your information

- at www.hra.nhs.uk/information-about-patients/
- the leaflet available from www.hra.nhs.uk/patientdataandresearch
- by asking one of the research team (see phone numbers below)
- by sending an email to the Data Protection Officer at RM. Email: dpo@rmh.nhs.uk.

#### **Contact numbers:**

#### GI

Royal Marsden NHS Foundation Trust, Sutton, Surrey

| Professor Cunningham | (Consultant) | 020 8661 3156 |
|----------------------|--------------|---------------|
| Dr Ian Chau | (Consultant) | 020 8661 3582 |
| Dr Sheela Rao | (Consultant) | 020 8661 3159 |
| Dr David Watkins | (Consultant) | 020 8661 3158 |
| Specialist Registrar | | 020 8642 6011 |
| Kennaway Ward | | 020 8661 3128 |
| West Wing | | 020 8661 6669 |
| On Call Registrar | (24 hours) | 020 8642 6011 |
| - | | |

| Research Nurse I | Name |
|------------------|------|

Contact Telephone No (9am – 5pm Mon – Fri) .....

CCR no: 5287 IRAS no: 282755

Version Date: 10th July 2020


| Rov | al Marsden | NHS | Foundation | Trust. | Fulham Road, | London |
|-----|------------|-----|------------|--------|--------------|--------|

| Professor Cunningham | (Consultant) | 020 7808 2123 |
|----------------------|--------------|---------------|
| Dr Ian Chau | (Consultant) | 020 8661 3582 |
| Dr Naureen Starling | (Consultant) | 020 7808 2123 |
| Senior Registrar | , | 020 7352 8171 |
| Burdett Coutts Ward | (24 hours) | 020 7808 2370 |
| On Call Registrar | (24 hours) | 020 7352 8171 |
| Research Nurse Name | | |

Contact Telephone No (9am – 5pm Mon – Fri) .....

#### Lymphoma

Royal Marsden NHS Foundation Trust, Sutton, Surrey

| Professor Cunningham | (Consultant) | 020 8661 3156 |
|----------------------|--------------|---------------|
| Dr Ian Chau | (Consultant) | 020 8661 3582 |
| Specialist Registrar | | 020 8642 6011 |
| Bud Flanagan West | | 020 8661 3144 |
| On Call Registrar | (24 hours) | 020 8642 6011 |
| West Wing | | 020 8661 6669 |
| Research Nurse Name | | |

Contact Telephone No (9am – 5pm Mon – Fri).....

Royal Marsden NHS Foundation Trust, Fulham Road, London

| Professor Cunningham | (Consultant) | 020 7808 2123 |
|----------------------|--------------|---------------|
| Dr Ian Chau | (Consultant) | 020 8661 3582 |
| Specialist Registrar | · | 020 7352 8171 |
| Wilson Ward | | 020 7808 2378 |
| On Call Registrar | (24 hours) | 020 7352 8171 |

Research Nurse Name .....

Contact Telephone No (9am – 5pm Mon – Fri).....

#### **Patient Advice and Liaison Service (PALS)**

Telephone: 0800 783 7176

Address: Royal Marsden NHS Foundation Trust, Downs Road, Sutton, SM2 5PT

CCR no: 5287 IRAS no: 282755

Version Date: 10<sup>th</sup> July 2020


### The ROYAL MARSDEN NHS Foundation Trust

GI & Lymphoma Unit Fulham Road, London SW3 6JJ: 020-7808-2153 Downs Road, Sutton SM2 5PT: 020-8661-3156

#### PATIENT CONSENT FORM (Page 1 of 2)

Cancer: Rapid Diagnostics and Immune assessment for SARS-CoV-2 (COVID-19) Arm A

Name of researcher: Dr Sheela Rao, Consultant Medical Oncologist.

Please initial each box to agree and sign at the bottom of the form.

| 1. | I confirm that I have read and understood the information sheet (CARDS Arm A v2.0 Dated: 10/07/2020) for this study and have had an opportunity to ask questions which have been answered to my satisfaction. |
|---|---|
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, and without my medical care or legal rights being affected. |
| 3. | I agree that relevant sections of any medical notes and data collected during the study may be looked at by responsible individuals at the Royal Marsden Hospital, the trial sponsor, and the regulatory authorities where it is relevant to my taking part in research. I give permission for these individuals to have access to my records. |
| 4. | I give my permission to transfer information relative to my medical history to be analysed in other ethically approved studies and/or collaborations. |
| 5. | I agree to researchers using my samples for the purposes listed in the information sheet. I understand that I am giving biological samples as a donation for research. |
| 6. | I agree to have blood, saliva, and throat/nose swab samples taken for research |

CONTINUE TO NEXT PAGE

CCR no: 5287 IRAS no: 282755

Version Date: 10<sup>th</sup> July 2020


#### PATIENT CONSENT FORM (Page 2 of 2)

### Cancer: Rapid Diagnostics and Immune assessment for SARS-CoV-2 (COVID-19) Arm A

When completed, 1 copy for patient, 1 original for researcher, 1 copy to be kept with case notes.